CLINICAL TRIAL: NCT03139305
Title: Effect of Prolonged (72 Hour) Glucagon Administration on Energy Expenditure in Healthy Obese Subjects
Acronym: GIO B
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TRIMDFH 954476
Record Dates: First submitted 2017-04-10; First posted 2017-05-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: glucagon
MeSH Terms: conditions — Obesity | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Glucagon Low Dose (Active Comparator)
  Interventions: Drug: Glucagon
- Glucagon High Dose (Active Comparator)
  Interventions: Drug: Glucagon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glucagon — Low dose intravenous infusion for 72 hours at 12.5 ng/kg/min
  Arms: Glucagon Low Dose
Drug: Glucagon — High dose intravenous infusion for 72 hours at 25 ng/kg/min
  Arms: Glucagon High Dose
Drug: Placebo — Intravenous infusion of saline for 72 hours
  Arms: Placebo

SUMMARY:
The main purpose of this study is to examine the effect of prolonged (72 hour) administration of glucagon compared to placebo on energy expenditure in healthy, non-diabetic, obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years, inclusive.
* Body Mass Index (BMI) ≥27 to ≤45 kg/m2 and body weight <450 lbs.
* Stable body weight for 3 months (self-reported loss/gain <5%).
* Judged to be non-diabetic per the American Diabetes Association guidelines:

  1. fasting plasma glucose <126 mg/dL [7.0 mmol/L] and
  2. HbA1c <6.5% [48 mmol/mol]) and
  3. in good health on the basis of medical history, physical examination (PE), electrocardiogram (ECG), and normal laboratory values obtained from Screening visit labs.
* Understands the procedures and agrees to participate in the study program by giving written informed consent, and is willing to comply with the trial restrictions.
* Willing to avoid alcohol consumption for 48 hours prior to the inpatient study visit.
* Willing to avoid consumption of caffeine and caffeinated beverages for 24 hours prior to the inpatient study visit.
* Willing to avoid strenuous physical activity for 72 hours prior to the inpatient study visit.

Exclusion Criteria

* Treatment with any medication known to significantly impact body weight or energy metabolism (e.g., weight loss medications, atypical antipsychotics) within 3 months prior to screening except for stable physiological hormone replacement therapy (i.e., thyroid hormone, estrogen).
* Treatment with a selective serotonin reuptake inhibitor, a medication for depression or apomorphine within one week prior to screening due to interaction with Zofran.
* History of bariatric surgery.
* Current liver, renal, pulmonary, cardiac, oncologic, metabolic, gastrointestinal, or hematologic disease which the Investigator believes is clinically significant, including:

  a. Liver disease or liver injury as indicated by abnormal liver function tests (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, serum bilirubin) >3 × upper limit of normal (ULN), or history of hepatic cirrhosis.
* Impaired renal function as indicated by an estimated glomerular filtration rate (eGFR) <60 mL/min or urine albumin-to-creatinine ratio >35 mg/mmol.
* Significant cardiovascular disease, including Class III or greater congestive heart failure (CHF), coronary artery disease, second degree or greater heart block, or clinically significant arrhythmias; baseline second degree or greater heart block or prolonged QT syndrome (QTc interval ≥470 msec); or any major cardiovascular event within the last 3 years (including myocardial infarction [MI], transient ischemic attack, cerebrovascular accident [CVA], angina, and hospitalization due to CHF,transient ischemic attack, and CVA).
* Metabolic, or other endocrine disorders, including diagnosis of type 1 or type 2 diabetes mellitus [HbA1c ≥6.5%]), inadequately treated hyperthyroidism (thyroid stimulating hormone [TSH] below normal range) or hypothyroidism (TSH >ULN <10 U/mL and symptomatic or TSH >10 U/mL), Cushing's disease/syndrome, Addison's disease, hypogonadism, or genetic disorders linked to obesity.
* History of irritable bowel disease, recurrent nausea, or vomiting.
* Anemia (hemoglobin <12 g/dL in males, <11 g/dL in females).
* History of dyslipidemia: Fasting triglycerides (TG) >500 mg/dL and low-density lipoproteins (LDL) >250 mg/dL.
* Self-reported history of infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
* History of recurrent sleep disturbances and/or prone to sleep disturbances based on lifestyle or employment (e.g., variable work schedule, overnight shift work, etc.).
* Diagnosis of sleep apnea with or without use of continuous positive airway pressure/BiPAP/AutoPAP.
* Major surgery within 3 months prior to screening.
* Blood donation within 4 weeks prior to screening.
* Participation in another investigational trial within 4 weeks prior to screening. The 4 week window will be derived from the date of the last trial medication and/or blood collection in a previous trial and/or adverse event (AE) related to trial drug screening of the current trial.
* Use of illicit drugs or nicotine-containing products within 3 months prior to screening.
* Poor intravenous (IV) access.
* Blood pressure <100/50 mmHg or ≥160/100 mmHg during screening.
* Heart rate ≥100 bpm during screening.
* Fasting plasma glucose <60 mg/dL or ≥126 mg/dL during screening.
* Female subjects who are, or intend to become, pregnant during the course of this study, are currently breastfeeding, or women of child-bearing potential (WOCBP) who refuse to use at least one method of birth control (oral contraceptives, intrauterine device, implanted or injectable contraceptives, abstinence).
* Translational Research Institute for Metabolism and Diabetes (TRI-MD) staff member or immediate relative of TRI-MD staff members directly involved
* History of any illness or condition that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Energy Expenditure | 24 hours
Effects of continuous IV infusion of glucagon versus placebo | 72 hours
  Overall well-being will be measured by administering a questionnaire with a scale from none to severe.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Smith, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arafat AM, Kaczmarek P, Skrzypski M, Pruszynska-Oszmalek E, Kolodziejski P, Szczepankiewicz D, Sassek M, Wojciechowicz T, Wiedenmann B, Pfeiffer AF, Nowak KW, Strowski MZ. Glucagon increases circulating fibroblast growth factor 21 independently of endogenous insulin levels: a novel mechanism of glucagon-stimulated lipolysis? Diabetologia. 2013 Mar;56(3):588-97. doi: 10.1007/s00125-012-2803-y. Epub 2012 Dec 22. PMID 23262585
- [Background] Astrup A, Rossner S, Van Gaal L, Rissanen A, Niskanen L, Al Hakim M, Madsen J, Rasmussen MF, Lean ME; NN8022-1807 Study Group. Effects of liraglutide in the treatment of obesity: a randomised, double-blind, placebo-controlled study. Lancet. 2009 Nov 7;374(9701):1606-16. doi: 10.1016/S0140-6736(09)61375-1. Epub 2009 Oct 23. PMID 19853906
- [Background] Calles-Escandon J. Insulin dissociates hepatic glucose cycling and glucagon-induced thermogenesis in man. Metabolism. 1994 Aug;43(8):1000-5. doi: 10.1016/0026-0495(94)90180-5. PMID 8052138
- [Background] Cegla J, Troke RC, Jones B, Tharakan G, Kenkre J, McCullough KA, Lim CT, Parvizi N, Hussein M, Chambers ES, Minnion J, Cuenco J, Ghatei MA, Meeran K, Tan TM, Bloom SR. Coinfusion of low-dose GLP-1 and glucagon in man results in a reduction in food intake. Diabetes. 2014 Nov;63(11):3711-20. doi: 10.2337/db14-0242. Epub 2014 Jun 17. PMID 24939425
- [Background] Cryer PE. Minireview: Glucagon in the pathogenesis of hypoglycemia and hyperglycemia in diabetes. Endocrinology. 2012 Mar;153(3):1039-48. doi: 10.1210/en.2011-1499. Epub 2011 Dec 13. PMID 22166985
- [Background] Flint A, Raben A, Rehfeld JF, Holst JJ, Astrup A. The effect of glucagon-like peptide-1 on energy expenditure and substrate metabolism in humans. Int J Obes Relat Metab Disord. 2000 Mar;24(3):288-98. doi: 10.1038/sj.ijo.0801126. PMID 10757621
- [Background] Kim J, Heshka S, Gallagher D, Kotler DP, Mayer L, Albu J, Shen W, Freda PU, Heymsfield SB. Intermuscular adipose tissue-free skeletal muscle mass: estimation by dual-energy X-ray absorptiometry in adults. J Appl Physiol (1985). 2004 Aug;97(2):655-60. doi: 10.1152/japplphysiol.00260.2004. Epub 2004 Apr 16. PMID 15090482
- [Background] Melzack R, Rosberger Z, Hollingsworth ML, Thirlwell M. New approaches to measuring nausea. CMAJ. 1985 Oct 15;133(8):755-8, 761. PMID 4042058
- [Background] Miyoshi H, Shulman GI, Peters EJ, Wolfe MH, Elahi D, Wolfe RR. Hormonal control of substrate cycling in humans. J Clin Invest. 1988 May;81(5):1545-55. doi: 10.1172/JCI113487. PMID 3284915
- [Background] Nair KS. Hyperglucagonemia increases resting metabolic rate in man during insulin deficiency. J Clin Endocrinol Metab. 1987 May;64(5):896-901. doi: 10.1210/jcem-64-5-896. PMID 2881943
- [Background] Salem V, Izzi-Engbeaya C, Coello C, Thomas DB, Chambers ES, Comninos AN, Buckley A, Win Z, Al-Nahhas A, Rabiner EA, Gunn RN, Budge H, Symonds ME, Bloom SR, Tan TM, Dhillo WS. Glucagon increases energy expenditure independently of brown adipose tissue activation in humans. Diabetes Obes Metab. 2016 Jan;18(1):72-81. doi: 10.1111/dom.12585. Epub 2015 Nov 20. PMID 26434748
- [Background] SCHULMAN JL, CARLETON JL, WHITNEY G, WHITEHORN JC. Effect of glucagon on food intake and body weight in man. J Appl Physiol. 1957 Nov;11(3):419-21. doi: 10.1152/jappl.1957.11.3.419. No abstract available. PMID 13480952
- [Background] Tan TM, Field BC, McCullough KA, Troke RC, Chambers ES, Salem V, Gonzalez Maffe J, Baynes KC, De Silva A, Viardot A, Alsafi A, Frost GS, Ghatei MA, Bloom SR. Coadministration of glucagon-like peptide-1 during glucagon infusion in humans results in increased energy expenditure and amelioration of hyperglycemia. Diabetes. 2013 Apr;62(4):1131-8. doi: 10.2337/db12-0797. Epub 2012 Dec 17. PMID 23248172
- [Derived] Whytock KL, Carnero EA, Vega RB, Tillner J, Bock C, Chivukula K, Yi F, Meyer C, Smith SR, Sparks LM. Prolonged Glucagon Infusion Does Not Affect Energy Expenditure in Individuals with Overweight/Obesity: A Randomized Trial. Obesity (Silver Spring). 2021 Jun;29(6):1003-1013. doi: 10.1002/oby.23141. PMID 34029448
- See also: Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org